CLINICAL TRIAL: NCT00568282
Title: Identification of Circulating Tumor Cells in the Peripheral Blood of Lung Cancer Patients (Old Title: Significance of CD44 and or Epithelial Specific Antigen Positive Cells in the Peripheral Blood of Lung Cancer Patients) (LUN0017)
Brief Title: Identification of Circulating Tumor Cells in the Peripheral Blood of Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-4086; 96710 (Other: Stanford University Alternate IRB Approval Number); LUN0017 (Other: Stanford University); 4086 (Other: Stanford IRB)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: phlebotomy — Standard of care
  Other Names: blood draw

SUMMARY:
The primary aim of this study is to determine whether we can identify human lung cancer tumor cells in the peripheral blood of lung cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether we can identify lung cancer cells circulating in the peripheral blood of lung cancer patients using cell surface markers found on cancer cells such as CD44 and epithelial specific antigen.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:Inclusion Criteria (Cases):

1. Advanced stage (IIIB with malignant effusion or IV) histologically or cytologically confirmed NSCLC
2. Patients must be newly diagnosed (untreated) or have evidence of disease progression at the time of sample collection
3. ability to sign informed consent
4. at least 18 years of age

Inclusion Criteria (Controls):

1. no known prior or active malignancy
2. ability to sign informed consent
3. at least 18 years of age Exclusion Criteria:1. history of any other cancer other than non-melanoma skin cancer within the last 5 years Exclusion Criteria:1. history of any other cancer other than non-melanoma skin cancer within the last 5 years

2. pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced stage NSCLC who are either newly diagnosed, or who have evidence of disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
to determine whether we can identify human lung cancer tumor cells in the peripheral blood of lung cancer patients using cell surface markers found on cancer cells. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. Wakelee, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States